CLINICAL TRIAL: NCT07323446
Title: 8-Week Double-Blind, Randomized Controlled Study of N-Acetylcysteine and Neuroimaging in Children Ages 6-12 With Emotional Dysregulation
Brief Title: The MIND Study: The MGH/MIT Investigation of NAC on Dysregulation
Acronym: MIND
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Janet Wozniak, MD, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P002315
Record Dates: First submitted 2025-12-11; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Emotional Dysregulation
Keywords: NAC; Emotional Dysregulation; Pediatric
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- N-Acetylcysteine (also known as NAC) (Experimental): Participants in the NAC arm will receive NAC in effervescent tablet form daily for 8 weeks . Participants will undergo neuroimaging before and after the 8-week treatment phase.
  Interventions:
  Drug: N-Acetylcysteine (NAC)
  Interventions: Drug: N-Acetyl Cysteine (NAC)
- Placebo (Placebo Comparator): Participants in the placebo arm will receive placebo (no active ingredients) in effervescent tablet form daily for 8 weeks. Participants will undergo neuroimaging before and after the 8-week treatment phase.
  Interventions: Drug: Placebo
- Control Group (No Intervention): Typically-developing controls will undergo neuroimaging twice (8 weeks apart) and will receive no intervention during the 8-week window.

INTERVENTIONS:
Drug: N-Acetyl Cysteine (NAC) — Participants in the NAC arm will receive NAC in effervescent tablet form daily for 8 weeks . Participants will undergo neuroimaging before and after the 8-week treatment phase.
  Arms: N-Acetylcysteine (also known as NAC)
Drug: Placebo — Participants in the placebo arm will receive placebo (no active ingredients) in effervescent tablet form daily for 8 weeks. Participants will undergo neuroimaging before and after the 8-week treatment phase.
  Arms: Placebo

SUMMARY:
This is a double-blind randomized controlled study. The study will last up to 16 weeks from the initial phone screen (it could take up to eight weeks to schedule and complete the initial screening process and schedule the 2 MRI visits). Once subjects have completed the screening process, they will begin the 8-week trial phase. Subjects will be assessed weekly throughout the study for efficacy and tolerability.

The investigators plan to recruit 80 participants with emotional dysregulation (ED) in the treatment arm. In addition, the investigators will aim to recruit 40age-, sex-, and parental-education matched participants without emotional dysregulation, and major psychopathology as Typically Developing (TD) control participants in the control arm.

Upon scheduling the baseline visit, only the emotional dysregulation (ED) participants will be randomized 1:1 to be exposed to NAC or placebo treatment for 8 weeks. Participants will complete baseline and post-treatment (endpoint) brain MRI acquisition. TD participants will complete the same screening and characterization process as the ED group and then will be invited to complete MRI eligibility screening and to be scanned twice, separated by an eight-week interval, but the TD will not complete the NAC treatment or receive a placebo. See Table 1 (Study Schema) for a complete list of characterization measures to be completed by each group.

DETAILED DESCRIPTION:
The investigators will enroll 120 subjects. Participants will be 80 children with emotion dysregulation, 6-12 years of age. In addition, the investigators will include 40 children without emotion dysregulation as healthy controls to provide a normative comparison group for neuroimaging analyses.

All subjects that enter the study will undergo standard screening and diagnostic procedures. Individuals who express interest in the study, either by responding to advertising or by giving a referring clinician explicit permission to be contacted for research, will be screened for eligibility by the study coordinator or a research assistant via phone. If the interested youth meet criteria for either the ED or TD group, the parent/guardian will be asked to complete the Child Behavior Checklist (CBCL) online via RedCap, a secure online data capture system.

The study coordinator will send a link to complete the CBCL electronically to the parent/guardian via email. An online consent statement will appear, prompting parents to indicate their agreement to participate in the online questionnaire portion of the study. If the parent/guardian indicates their agreement, the data capture system will proceed to the CBCL.

After completing the CBCL, eligible participants based on inclusion and exclusion criteria will either be assigned to the ED or TD group. Eligible participants will be scheduled to speak with a study clinician via phone or secure Zoom call to obtain informed consent prior to completing further screening and baseline study procedures.

Written informed consent will be obtained from subjects' parent/guardian prior to initiation of the study protocol. Subjects aged 7 and older will sign age-appropriate assent forms. The study subjects and their parent may take as much time as they feel necessary to consider their participation in the study as well as consult with their family members or physician. Subjects may remain on most current treatments while participating in this study. Participation in this study is voluntary, and subjects may withdraw from the study at any time.

Informed consent will be obtained virtually. Study staff will send the consent form and assent form (when applicable) to subjects in PDF form ready for Adobe eSignature via email with a brief statement explaining why they are receiving this form and further instructions. Study staff will schedule a time for the subject and their parent(s)/guardian to meet with a study clinician via phone or secure Zoom to complete consent. For the ED group, the study clinician will have a conversation over the phone or Zoom with the subject and their parent(s)/guardian to obtain consent in the usual fashion: review the consent form, review inclusion and exclusion criteria, review risks and benefits of the study, review alternatives to participation, and answer any questions subjects and their parent(s)/guardian may have. If the subject and their parent(s)/guardian decide to participate, they will sign the consent form and assent form (when applicable) using Adobe eSignature. The study clinician will also sign the consent form using Adobe eSignature prior to beginning any study procedures. Subjects will be sent a copy of the signed form by email for their records. For the TD group, the same procedure will be followed but will be completed by the clinical research coordinator.

STUDY PROCEDURES

This will be an 8-week, double-blind randomized controlled study of NAC in the treatment of emotional dysregulation in children and adolescents. Subjects will include youth ages 6-12 years old. The primary outcome measures will be improvement in manic symptoms as measured by the Young Mania Rating Scale (YMRS) and improvement in depressive symptoms as measured by the Child Depression Rating Scale (CDRS).

The main outcome measures will be GSH levels in participants pre- and post- treatment as well as the Young Mania Rating Scale (YMRS) and the Children's Depression Rating Scale (CDRS).

The Child Behavior Checklist (CBCL) will be collected during pre-screening procedures and at post-treatment. The CBCL is used for inclusion in the study and a measure of psychiatric symptoms across multiple domains.

Pre-Screening Parents/guardians who inquire about having their child participate in this study and who provide explicit permission to be contacted for research will be contacted by a member of study staff to be screened by phone for inclusion and exclusion criteria. If a child may be eligible, detailed contact information will be collected. If a parent/guardian gives consent and their child gives assent to participate at the following screening/baseline visit, information regarding the child's medical, health, and psychiatric history that was collected in the phone screen will be stored securely with the other data that is collected during study participation. If the child does not enroll in the study for any reason, this information will be de-identified.

Potential subjects who meet eligibility criteria during the phone screen will be asked to complete the CBCL electronically via RedCap. The study coordinator will send the parent/guardian a link to complete the CBCL electronically via encrypted email, unless the parent/guardian has explicitly requested to receive email correspondence without encryption. The links will be unique to the subject, preventing subjects and their parent/guardian from accessing any other data stored on the password-protected database. This link will direct the parent/guardian to a page with a written consent statement about this portion of the research. The parent/guardian will then be asked to indicate their agreement to continue with the CBCL by clicking the appropriate button, providing electronic consent to participate in the online questionnaire. If the parent agrees to complete the CBCL, they will be directed to the online questionnaire.

The CBCL should take approximately 20 minutes to complete. If the potential subject meets eligibility criteria based on the CBCL scores, the coordinator will contact the parent/guardian to schedule a virtual screening/baseline visit with a study clinician. If the parent/guardian gives consent and their child gives assent to participate at the following screening/baseline visit, the parent/guardian's responses to the online CBCL questionnaire completed during pre-screening will be stored securely with the other data that is collected during study participation. If the child does not enroll in the study for any reason, this information will be de-identified.

Baseline Visit

After the consent/assent form is signed, the investigators will do the following:

Have the parent/guardian complete questionnaires through REDCap prior to the visit (study coordinator will email link ahead of time) regarding:

* Current medications
* Demographic details
* Parent-Young Mania Rating Scale (P-YMRS)
* Social Responsiveness Scale (SRS) questionnaire (ED only)
* Parent-completed Children's Depression Rating Scale (CDRS) (ED only)
* The Modified Overt Aggression Scale (MOAS) (ED only)
* MIT MRI Metal Safety Screening Form

A study clinician will review this information and meet with parent/guardian and child during a virtual visit over Zoom. In this visit, the clinician will:

* Review current medications (ED only)
* Complete the Columbia Suicide Severity Rating Scale (C-SSRS) assessing past and current suicidality and self-harmful behaviors
* Record baseline severity scores of Clinical Global Impression (severity scores) for mania, depression and overall bipolar disorder (ED only)
* Complete the Young Mania Rating Scale (YMRS) to assess manic symptoms

All assessments and scales will be completed via REDCap.

The study coordinator will also complete a phone call with the ED subjects and their parent(s)/guardian on the same day as the tele-visit with the study clinician in order to complete the following procedures. Parents/guardians will be asked to self-report height and weight of their child. It will be noted that these measurements were provided by a parent/guardian report rather than study staff measurement.

The investigators expect most homes will have measures for weight and height and will request this information at the first visit. However, if this is not the case, the investigators can provide measuring tools. Proper safety procedures will be reviewed with subjects and parents, including the use of 911 for emergencies and how to contact the study clinician or covering clinician 24/7. Those subjects who terminate study participation before the completion of the study will be asked to complete all tasks scheduled to take place on the final study visit at the time of study discontinuation.

Randomization Randomization to NAC or placebo will occur once a subject is scheduled for a baseline visit when the clinical trials pharmacy will be given a subject name that the pharmacy will associate with a number identifier. Randomization lists stratified by gender and age will be generated by our statistician and utilized by the MGH Clinical Trials Pharmacy. The investigators have extensive experience maintaining blinding, wherein the investigators have our central Mass General Hospital Clinical Trials Pharmacy serve as the only part of the greater trial team that is aware of the assignment to active or placebo during study participation. The trials pharmacy will receive products identified by the sponsor as active or placebo fill package these products with unique identifiers, maintain the placebo-active ratio, and maintain blinding until study completion. For the purpose of the final analysis, the official clinical database will not be unblinded until medical/scientific review has been completed, protocol violators have been identified (if appropriate), and data collection has been declared complete. In the extreme event where subject safety will be compromised by maintaining the blind, eg. an adverse event where treatment is dependent on knowing if they were on active or placebo medication, the investigators will unblind the status of the subject's study agent, following emergency protocols in place in our department and institution.

Dosing Active and placebo study treatment will be purchased from BioAdvantex. ED subjects will receive effervescent tablets of NAC. Subjects will receive 1800mg (2 900mg tablets) of NAC daily or a matched placebo. This dosing was selected based on a previous successful open-label trials of NAC in youth (Wozniak, DiSalvo et al. 2022). The child will take the study drug (or placebo) by drinking a tablet dissolved in a liquid, either twice a day or once a day according to personal preference, for the entire study.

Remote Study Medication Dispensation Study medication will be shipped by BioAdvantex to MGH Clinical Trials Pharmacy (CTP) where it will be stored and dispensed. Randomization lists stratified by gender and age will be generated by our statistician and utilized by the MGH Clinical Trials Pharmacy. Study staff will pick up the study medication that is assigned to each participant from the MGH CTP, remaining blinded to whether it is an active or placebo product, and send it via courier mail service directly to the participant's home address, only if the participants reside in the state of Massachusetts. Staff will be trained to follow all guidelines elaborated by the MGH CTP and Drug Enforcement Agency in this process. The study medication will be ordered and shipped following the baseline study visit, with sufficient supply to cover participation for all 8 weeks. An additional week of study treatment will be sent to cover any time between the end of Week 8 and when the final MRI scan is scheduled. Patients will remain on study drug until the follow up visit after the EP MRI and thus overage is being provided to get them through to that visit. A member of the study staff will contact the participant with the estimated date and time of the prescription delivery as well as the tracking number to ensure proper retrieval.

No study medication will be shipped to participants outside the state of Massachusetts. Participants residing outside of the state of Massachusetts will pick up the study medication at MGH.

Close contact by the study team with the participants to monitor medication intake will continue throughout the study. Individuals will be given clear instructions to adhere to the agreed-upon dosing schedule between study visits, must keep the study agent in a safe place where others would not take it in error, must not divert any study agent, and must return study medication to the investigators at the end of the study. Per standard research procedure, the study clinician will record reported medication compliance in the applicable RedCap Note.

After the completion of study participation, the participant will send the leftover study medication to the study coordinator. Participants will be provided with FedEx shipping materials to return any remaining study medication. The study coordinator will complete a thorough tablet count at that time and maintain the study medication until it can be returned to MGH and discarded per the MGH CTP destruction policy.

Concomitant Medications A detailed past and present treatment history will be taken as part of initial evaluation. Taking NAC with other medications or supplements may change how the study treatment(s) or other medications or supplements work. Study clinicians will monitor concomitant medications and their potential interactions with the study treatment(s) or impact on our outcome measures.

Patients who are partially responding to current psychotropic medication yet continue to have symptoms of emotional dysregulation, mania, or depression will be permitted to continue on their current regimen, provided the patient's regimen remains the same throughout the study. Patients treated with these medications must be on a stable dose for at least two weeks prior to study entry. No new medications (except for the use of the benzodiazepine lorazepam listed below) or alterations to the current regimen may be initiated throughout the duration of study participation.

The use of the benzodiazepine lorazepam is permitted during the study. Patients may not exceed a dosage of 2mg lorazepam per day and lorazepam is permitted for a maximum of 3 days during the study. Any greater need for lorazepam will be considered evidence of poor treatment response and grounds for drop from the study.

Non-pharmacological treatments such as individual, family or group therapy will be allowed if they were in place before the patient joined the study. The patient's therapy regimen must remain the same throughout the study. No new non-pharmacological treatments may be initiated after study participation has begun.

Pre- and Post-Treatment Scanning Visits MRI scanning will be performed at the A.A. Martinos Imaging Center at MIT (43 Vassar Street, Cambridge, MA 02139). All participants (children with and without emotion dysregulation) will complete two scanning visits. The first scanning visit, or the pre-treatment scanning visit, will take place +/- 2 days from the screening/baseline visit. The second visit, or the post-treatment scanning visit, will take place during Week 8 while the subject is still taking the treatment. This will take place within 5 business days of the end of Week 8. If a participant terminates the study for any reason after week 2 and before week 8, the post-treatment scan can be conducted before the completion of the full trial. If a participant stops taking NAC before the final scan, no more than a 48-hour gap between the last NAC dose and the scan will occur.

Weekly Visits (Weeks 1 through 8)- ED group only ED subjects will receive study treatment as indicated by a double-blind placebo controlled RCT schedule.

Study visits will occur at 14-day intervals but have a visit window of +/- 2 days to facilitate scheduling. All visits will occur via tele-psychiatry virtual visit platform.

On weeks when there is no scheduled study visit with the clinician, the study staff will call to to record medication compliance and tolerability, inform and schedule clinician visit to address concerns.

Each week, in addition to the tele-visit or check in call, parents will respond in REDCap via email link to:

* Indicate adherence to study treatment and # and times of missed dosing
* List new concomitant medications or treatment
* Complete parent-completed scales regarding symptoms of emotional dysregulation, mania, and depression (P-YMRS, CDRS and MOAS)

Every other week, during the tele-visit, the study clinician will:

* Complete the Columbia Suicide Severity Rating Scale (C-SSRS)
* Ask the parents/guardians further questions about their child's symptoms of emotional dysregulation completing Clinical Global Impression scales (severity and improvement) for mania, depression and overall bipolar disorder
* Record any side effects or adverse events
* Review and confirm parent recorded new concomitant medications or treatment
* Review and confirm parent recorded adherence to study treatments recording # of missed doses

At the week 8 (or final) study visit, the email link sent to parents will also have them:

* List current weight
* Complete the SRS questionnaire
* Complete the CBCL questionnaire

Study Discontinuation Subjects may drop at any time due to patient preference, physician decision, need for psychiatric hospitalization, or a poor response to treatment. Poor response to treatment will be measured by a CGI-bipolar score that is 2 points higher (more severe) than baseline for 2 weeks in a row or a P-YMRS score that is 30% higher than baseline for 2 weeks in a row only if the P-YMRS is in a clinically significant range of >15, which may lead to drop from the study as determined by the clinician. Initial and emergent suicidality will be assessed weekly through administration of the Columbia Suicide Severity Rating Scale (C-SSRS). Subjects scoring 4 or higher will be dropped from the study. If emergent suicidality were to occur during the course of the study, the supervising clinician will then directly assess the level of risk and take the appropriate action (including contacting treatment providers, working on a safety plan, arranging for emergency evaluation via an ER, calling 911, etc.) The clinician will document the actions taken, and it will be noted in the participant's file. In addition, drop from study will occur at clinician discretion for worsening of clinical course, non-compliance with treatment, or inability to tolerate study treatment.

Subjects who fail to keep study appointments or are non-compliant (less than 70% compliance for two weeks or longer) may be dropped from the study.

If a subject becomes pregnant or is found to be abusing substances during the study, he or she will be discontinued from the study and given a referral for local treatment.

If a subject would like us to forward their clinical history to his/her primary care physician, or a new clinician, the investigators will forward any pertinent information if an appropriate signed release of information is provided. If a subject who has come from the clinic of the investigator happens to drop out of the study, he or she will return to his or her treating physician.

ELIGIBILITY:
Inclusion Criteria:

- Emotional Dysregulation Group

1. Male or female subjects, 6-12 years of age.
2. Current symptoms of emotional dysregulation as indicated by combined T-scores on the Child Behavior Checklist > 180 on the Anxiety/Depression + Aggression + Attention subscales.
3. Score 15 or above on the clinician YMRS
4. Subjects and their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
5. Subjects and their legal representative must be considered reliable.
6. Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must provide written consent and the subject must provide written assent.
7. Subject must have access to a computer with a camera, speaker, microphone, and internet connection.
8. Subject must be willing to refrain from treatment changes during the study protocol.

Typically Developing Control Group

1. Age-, sex-matched with ED participants.
2. No significant traits of ED as screened by parent and clinician YMRS both under scores of 6
3. No previous psychiatric history as confirmed by clinician interview
4. No significant psychopathology as screened on the CBCL (Subdomain T-scores <60).
5. Participant weight is above the 5th percentile and below the 95th percentile, per CDC child BMI categories (https://www.cdc.gov/obesity/basics/childhood-defining.html)

Exclusion Criteria:

1. Investigator and his/her immediate family (defined as the investigator's spouse, parent, child, grandparent, or grandchild).
2. Serious or unstable illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
3. History of bleeding diathesis, including those with von Willebrand disease.
4. Uncorrected hypothyroidism or hyperthyroidism.
5. History of sensitivity to N-acetylcysteine, a history of intolerance to N-acetylcysteine or a non-responder after 2 months of treatment at adequate doses as determined by the clinician.
6. Severe allergies or multiple adverse drug reactions.
7. Current or past history of seizures.
8. DSM-IV substance use, abuse, or dependence
9. Any concomitant medication with primary central nervous system activity other than specified in the Concomitant Medication portion of the protocol.
10. Current diagnosis of schizophrenia or psychosis.
11. Females who have started menstruating.
12. Pregnant or nursing.
13. Judged to clinically be at serious suicidal risk or C-SSRS score ≥ 4.
14. History of intellectual disability as reported by parent

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change in the Clinician-Young Mania Rating Scale (C-YMRS) Score | Baseline to Endpoint (Week 8)
  The YMRS consists of 11 items rated on a scale from 0 (symptoms not present) to 4 (symptoms extremely severe). It is used to assess manic symptoms. Scores from each item are summed to obtain the total YMRS score. The YMRS score ranges from 0-60. A higher score means a higher manic state. Questions are asked about the last week. This scale is generally accepted as the main outcome measure in studies of pediatric bipolar disorder and is linked directly to the core symptoms of mania.
Mean Change in the Clinical Global Impression (CGI) scale for mania, depression, and bipolar disorder. | Baseline to Endpoint (Week 8)
  The CGI is a measure of illness severity adapted for specific disorders. It allows rating of mania, depression, and overall bipolar disorder illness, as well as other conditions frequently comorbid with bipolar disorder.
  The severity score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The improvement score ranges from 1 (very much improved) to 7 (very much worse).
  Collected at the baseline visit, weeks 2, 4 and 6, and at endpoint as an accepted measure of clinician rated improvement to assess the impact of treatment on bipolar disorder and other comorbid conditions.
Change from baseline to endpoint in the clinician measure Children's Depression Rating Scale (CDRS) | Baseline to Endpoint (Week 8)
  The CDRS (Poznanski, Freeman et al. 1985) is modeled after the Hamilton Depression Rating Scale for adults, but includes questions relevant to youth, such as questions about school, family and peer functioning.
  This is a clinician-rated instrument with 17 items scored on a 1 to 5 or 1 to 7 scale. A rating of 1 indicates normal, thus the minimum score is 17. The maximum score is 113. Scores of 20-30 suggest borderline depression. Scores of 40-60 indicate moderate depression.
  This scale is generally accepted as the main outcome in studies assessing childhood depression and is linked directly to the core symptoms of depression.
  Collected at baseline visit, weeks 2, 4 and 6, and at endpoint.

SECONDARY OUTCOMES:
Mean Change in Child Behavior Checklist (CBCL) scores | Baseline to Endpoint (Week 8)
  The CBCL (Achenbach 2000) is a standardized assessment of child behavior problems and social competence. Due to its extensive use and available norms, it provides us with an effective method of comparing our sample with others in the literature.
  The CBCL records, in standardized format, the behavioral problems and competencies of children aged 4 to 18, as reported by their parents or parent- surrogates.
  The CBCL is scored on the recently revised social competence and behavior problem scales of the Child Behavior Profile. A T-score above 70 is considered to be a clinically meaningful indicator of childhood psychopathology.
  Administered during pre-screening procedures as part of inclusionary criteria as well as at post-treatment completion.
Mean Change in Social Responsiveness Scale (SRS) Scores | Baseline to Endpoint (Week 8)
  The SRS is a 65-item rating scale completed by the parent or guardian. This scale measures the severity of autism spectrum symptoms as they occur in natural social settings.
  Collected at screening and endpoint visits as assessment of symptoms and capacities associated with social interaction.
Mean Change in the Parent-Young Mania Rating Scale (P-YMRS) Score | Baseline to Endpoint (Week 8)
  The P-YMRS (Young, 1978) consists of 11 items rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe).
  Items 5, 6, 8, and 9 are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). These items assess irritability, speech, content, and disruptive/aggressive behavior) and are given extra weight in the overall score.
  The YMRS score ranges from 0-60. Questions are asked about the last week. This scale is generally accepted as the main outcome measure in studies of pediatric bipolar disorder and is linked directly to the core symptoms of mania.
  Collected at the screening visit, baseline visit, at each of the weekly visits, and at endpoint to assess the impact of treatment on manic symptoms
Mean Change in the Children's Depression Rating Scale-Parent (CDRS-P) Score | Baseline to Endpoint (Week 8)
  Scale for adults, but includes questions relevant to youth, such as questions about school, family and peer functioning.
  This is a parent-rated instrument with 17 items scored on a 1 to 5 or 1 to 7 scale. A rating of 1 indicates normal, thus the minimum score is 17. The maximum score is 113. Scores of 20-30 suggest borderline depression. Scores of 40-60 indicate moderate depression.
  This scale is generally accepted as the main outcome in studies assessing childhood depression and is linked directly to the core symptoms of depression.
  Collected weekly
Mean Change in the Modified Overt Aggression Scale (MOAS)- Parent | Baseline to Endpoint (Week 8)
  The MOAS is a 4-item rating scale completed by the parent or guardian. This scale measures aggressive behavior over the previous week.
  Collected weekly as assessment of change in aggression throughout the 8-week study

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts Institute of Technology, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: No